CLINICAL TRIAL: NCT00935805
Title: ANALYSIS OF THE EFFECTIVENESS OF A STAGED MANAGEMENT PROGRAM AIMED AT CONTROLLING BLOOD PRESSURE AND BLOOD GLUCOSE OF TYPE 2 DIABETIC PATIENTS USING EXCLUSIVELY THE RESOURCES AVAILABLE IN A PRIMARY CARE SETTING IN BRAZIL
Brief Title: Glycemic And Blood Pressure Control In Type 2 Diabetes, In A Primary Care Unit: A Staged Management Strategy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: 06260
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus; Arterial Hypertension
Keywords: Diabetes Mellitus; Arterial Hypertension; Treatment; Primary Care
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Metformin; Glyburide; Insulin, Isophane; Hydrochlorothiazide; Propranolol; Captopril; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: 124 patients attending the primary care unit included after formal consent.
  Interventions: Drug: Metformin; Drug: Glybenclamide; Drug: NPH insulin; Drug: Hydrochlorothiazide; Drug: Propranolol; Drug: Captopril; Drug: Amlodipine

INTERVENTIONS:
Drug: Metformin — 850 mg TID
  Other Names: Initial drug added to non-pharmacological measures
Drug: Glybenclamide — 10 mg BID
  Other Names: Second oral agent to be added
Drug: NPH insulin — Variable SC dose
  Other Names: Insulin added to or substituted for OA
Drug: Hydrochlorothiazide — 25 mg QD introduced as initial therapy for hypertension
  Other Names: Inital RX for hypertension
Drug: Propranolol — 40 mg BID
  Other Names: Introduced if diuretic + captopril do not control BP
Drug: Captopril — 50 mg TID
  Other Names: Added to hydrochlorothiazide if BP not attained
Drug: Amlodipine — 10 mg QD
  Other Names: Added to previous if BP control BP not satisfactory

SUMMARY:
The aim of this study is to to analyze if it is possible to reach the goals of HbA1c <7.0% and blood pressure <= 130/80 mm Hg in a cohort of patients with type 2 diabetes attending a primary care unit, using ony those resources available at the unit, and provided by the Brazilian National Health System. It is an open label, observational study, with a duration of 4-6 years. Patients attending a primary care outpatient facility will be sequentially included in the study provided they give consent. They will be followed on a monthly basis by a team of physicians and nurses. Glucose, A1c, Blood PRessure will be the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (WHO)

Exclusion Criteria:

* Terminal disease (renal, cancer, heart failure)

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients attending a primary care outpatient facility
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2006-07; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin A1c | 3 months
Blood pressure | 1 month

SECONDARY OUTCOMES:
24 hr blood glucose profile | once
Fasting blood glucose | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rogerio Friedman, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Jorge L Gross, MD, PhD, Study Chair — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil